CLINICAL TRIAL: NCT03347890
Title: Central Nervous System Effects of Liraglutide® 3.0 mg on Reward Mechanisms in Obese Patients Without Diabetes, in Relation to Food Addiction. A Randomized, Single-centre, Double-blind, Placebo Controlled Clinical Trial.
Brief Title: Reward Mechanisms in Obesity
Acronym: LIRAOB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zoltan Pataky (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Zoltan Pataky, MD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-01085; U1111-1194-9675 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2017-11-12; First posted 2017-11-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: GLP-1; fMRI
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Randomized, single-centre, double-blind, placebo controlled, parallel group, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide 3.0 mg (Experimental): 35 obese patient will be evaluated at baseline and at 16-week (end of study) after daily subcutaneous injections of Saxenda® (liraglutide 3.0 mg).
  Interventions: Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml or Placebo
- Placebo (Placebo Comparator): 35 obese patient will be evaluated at baseline and at 16-week (end of study) after daily subcutaneous injections of Placebo by pen injector.
  Interventions: Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml or Placebo

INTERVENTIONS:
Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml or Placebo — Patients will be evaluated at baseline and at 16-week (end of study) after daily subcutaneous injections of Saxenda® (liraglutide 3.0 mg) or Placebo by pen injector.

SUMMARY:
The study aims to investigate the effects of 3.0 mg of liraglutide on reward brain circuits in human obesity and to better understand its effects on weight loss (in patients without diabetes).

According to the study protocol, 70 obese patient will be evaluated at baseline and at 16-week (end of study) after daily subcutaneous injections of Saxenda® (liraglutide 3.0 mg) or Placebo by pen injector.

All participants will first undergo a functional Magnetic Resonance Imaging (fMRI) session while being presented with gustatory stimuli. Second, participants will complete behavioural tasks (i.e., liking versus wanting, in the scanner) and questionnaires aiming at teasing apart reward mechanisms and emotional skills (e.g., emotional regulation ability) associated with food intake. Third, metabolic parameters and hormones involved in appetite regulation will be assessed and studied in relation to fMRI.

These measurements will be repeated after 16 weeks in obese individuals. The control group of normal body weight individuals will be evaluated once at Baseline.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 and < 40 kg/m2
* right-handed
* current non-smokers
* with stable body weight (<5% reported change during the previous 3 months)

Exclusion Criteria:

* History of any psychiatric, neurological, cardiovascular, renal or liver disease, malignancies, type 1 and type 2 diabetes mellitus
* use of centrally acting medication, glucocorticoides, insulin, orlistat
* any substance abuse
* food allergies
* deficits of smell and taste
* history of pancreatitis
* family or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma
* pregnancy
* contraindications for fMRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change of Bold Oxygenation Level Dependent (BOLD) signal (%) in brain regions involved in the reward system | 16 weeks
  Bold changes in striatum, amygdala, insula, orbitofrontal complex as detected by fMRI in from baseline to 16-week follow-up

SECONDARY OUTCOMES:
change of body weight | 16 weeks
  Weight measurement (kg)
changes in waist circumference | 16 weeks
  waist circumference measurement (cm)
changes in fasting blood sugar | 16 weeks
  fasting glycaemia measurement (mmol/l)
changes in glucagon | 16 weeks
  glucagon measurement (pmol/l)
changes in ghrelin | 16 weeks
  ghrelin measurement (mg/dl)
changes in leptin | 16 weeks
  leptin measurement (ng/ml)
changes in obestatin | 16 weeks
  obestatin measurement (ng/ml)
changes in reelin | 16 weeks
  reelin measurement (ng/microL)
changes in endocannabinoids | 16 weeks
  measurement of anandamide (AEA), 2-arachidonoylglycerol (2-AG), N-palmitoylethanolamide (PEA), N-oleoylethanolamide (OEA); ng/ml for all
changes in insulin | 16 weeks
  fasting insulinaemia measurement (mUI/l)
change in food addiction score | 16 weeks
  Assessment by YFAS V.2 questionnaire, 25 questions, total score is reported
change in liking | 16 weeks
  Assessment by Pavlovian-Instrumental Transfer (PIT) test during fMRI scanning. Participants will taste the milkshake and tasteless solutions and asked to rate them based on how much they liked tasting the stimulus on a visual analogue scale (ranging from 1 "not at all" to 100 "extremely").
change in wanting | 16 weeks
  Assessment by Pavlovian-Instrumental Transfer (PIT) test during fMRI scanning. We will measure the mobilized effort (using a handgrip) the participants mobilized to be delivered with the milkshake.
change in emotional regulation abilities | 16 weeks
  Assessed by an emotional regulation task. Subjects will be presented with neutral, positive, negative, and mixed emotional feelings film clips and asked to either attend naturally or decrease their emotional reactions. The clips will be rated on amusement and repulsion scales on a 6-point scale. Based on these ratings, we will calculate a mixed feelings coefficient.
BOLD in brain regions involved in the reward system | baseline comparison
  BOLD (%) in striatum, amygdala, insula, orbitofrontal complex as detected by fMRI in the obese groups at baseline in comparison to normal body weight controls

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Pataky, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No